CLINICAL TRIAL: NCT04185337
Title: The Role of Ultrasound-Guided Photoacoustic Imaging in Detection of Metastases in Inguinal Lymph Nodes
Brief Title: Ultrasound-Guided Photoacoustic Imaging for the Detection of Metastases in Inguinal Lymph Nodes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0461; NCI-2019-07316 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0461 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Biopsy, Fine-Needle; Sentinel Lymph Node Biopsy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (ultrasound, ultrasound-guided PAI, FNA, biopsy) (Experimental): Patients undergo standard of care ultrasound of the lymph nodes, then undergo ultrasound-guided PAI over 3-5 minutes. Patients then undergo standard of care ultrasound-guided FNA or biopsy a suspicious lymph node.
  Interventions: Procedure: Fine-Needle Aspiration; Procedure: Lymph Node Biopsy; Procedure: Photoacoustic Imaging; Procedure: Ultrasound; Device: Multispectral optoacoustic tomography (MSOT) acuity instrument

INTERVENTIONS:
Procedure: Fine-Needle Aspiration — Undergo ultrasound-guided FNA
  Other Names: Aspirate, Fine Needle; Fine Needle Aspiration; fine-needle aspiration biopsy; FNA; FNA biopsy
Procedure: Lymph Node Biopsy — Undergo ultrasound-guided lymph node biopsy
  Other Names: Biopsy of Lymph Node
Procedure: Photoacoustic Imaging — Undergo ultrasound-guided PAI
Procedure: Ultrasound — Undergo ultrasound
Device: Multispectral optoacoustic tomography (MSOT) acuity instrument — Use multispectral optoacoustic tomography (MSOT) acuity instrument

SUMMARY:
This early phase I trial studies how well ultrasound-guided photoacoustic imaging works in telling the difference between healthy and cancerous inguinal (groin) lymph nodes and how well it can detect certain features of lymph nodes, including size and shape in patients with cancer. Ultrasound-guided photoacoustic is a non-invasive imaging method that can detect and display characteristics of lymph nodes based on the level of oxygen in the cells. This imaging method may provide more accurate tumor staging and prevent unnecessary surgical interventions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the mean difference in oxygen saturation (%sO2) between healthy and malignant inguinal lymph nodes using ultrasound-guided photoacoustic imaging (PAI) in cancer patients.

SECONDARY OBJECTIVE:

I. To examine the role of ultrasound-guided PAI in detecting metastases in the inguinal lymph nodes and ultrasound features of lymph nodes such as the size, shape of the lymph nodes.

OUTLINE:

Patients undergo standard of care ultrasound of the lymph nodes, then undergo ultrasound-guided PAI over 3-5 minutes. Patients then undergo standard of care ultrasound-guided fine needle aspiration (FNA) or biopsy a suspicious lymph node.

After completion of study, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven primary malignancy
* Suspicious inguinal lymph nodes for metastasis on a conventional imaging modality
* Scheduled to undergo ultrasound-guided fine needle aspiration cytology or biopsy

Exclusion Criteria:

* Melanoma patients, since the melanocytes may have a "masking effect"
* The deeper inguinal lymph nodes (3-5 cm deep) and smaller (< 1 cm in short axis) in dimensions will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Difference between background oxygen saturation (%sO2) and nodal %sO2 | Up to 3 months
  For each suspicious lymph node, a %sO2 throughout the entire lymph node volume will be obtained. The %sO2 from the tissue immediately surrounding each lymph node will also be calculated to account for variations in background %sO2. The tumor status will be confirmed with ex vivo histopathology. Will scan normal lymph nodes in the same or contralateral inguinal region and will use as controls. Data will be analyzed once the benignities of these lymph nodes are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Priya R Bhosale, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04185337/ICF_000.pdf